CLINICAL TRIAL: NCT03515564
Title: Targeting Trauma-Related Disorders With Arts and Movement Therapies
Brief Title: Arts and Movement Therapies for Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Arash Javanbakht, Director of Stress, Trauma, and Anxiety Research Clinic, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1706000635
Record Dates: First submitted 2018-04-11; First posted 2018-05-03 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: PTSD; Depression; Anxiety; Stress; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Wounds and Injuries | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative therapy (Experimental): Dance/Movement Therapy, Art Therapy, Mindful Yoga
  60 minutes once weekly for 8 weeks
  Interventions: Behavioral: Dance/Movement Therapy, Art Therapy, Mindful Yoga
- No Intervention (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: Dance/Movement Therapy, Art Therapy, Mindful Yoga — Utilizing deep breathing, exercise modalities, and social support in all settings
  Arms: Alternative therapy

SUMMARY:
The current goal of this project is to subjectively and objectively assess the efficacy of arts and movement interventions--including dance/movement therapy, art therapy and mindful yoga for youth and adults exposed to trauma, including families resettled as refugees and families in high-risk, low-resource environments. The overarching aim is to measure the changes over time in self-reported symptoms of posttraumatic stress disorder, anxiety disorder(s), depression, and somatic symptoms, as well as changes in biological substrates representing pathophysiological processes involved in responses to stress, trauma, and the aforementioned disorders. These biological substrates include inflammatory proteins and the stress hormone cortisol. We hypothesize that given the emotional and physical components of arts and movement therapies, which are implemented in group settings and confer life-long coping skills to participants, participation in arts and movement therapies will result in reduction of self-reported severity of psyciatric symptoms and improved physiology.

COVID-19: In March, the COVID-19 pandemic caused in person research to be halted in order to be in adherence to the stay at home order for the State of Michigan. The IRB overseeing the present project approved an amendment to allow data to be collected online via phone or email, based on participant preference, with a new consent form for this new method of data collection. Following this approval, we migrated our programming to virtual formats and began to serve both refugee commuities as well as school-aged youth with the intervention program and obtained consent followed by data from participants as part of this study. We have pivoted towards also looking at the benefits of creative arts and movement based interventions in reducing COVID-related distress, as well as building resilience.

By collecting psychological and biomarker data the investigators seek concrete scientific evidence supporting these non-pharmacological, cost effective, and accessible programs as reliable treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children and adults ages 7-65
* Willing and able to consent, or with at least one parent willing and able to provide consent for minors under age 18

Exclusion Criteria:

* Adults who are unable or unwilling to consent, or children whose parent do not consent
* Wardens of the Court

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms (children) | 8 weeks
  Evaluation of PTSD related symptoms. UCLA Trauma Questionnaire administered to children. 33 items ranked from 0-4, with 0 = none of the time to 4 = most of the time. Scores can be summed for a composite score, with a maximum of 132 and a minimum of 0, or determination of PTSD criteria met utilizing responses to individual questions.

SECONDARY OUTCOMES:
PTSD symptoms (adults) | 8 weeks
  PCL-c for DSM V (Post-traumatic stress disorder checklist for civilians). 20 questions ranked from 0 to 4 for "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." Maximum score = 80, minimum score = 0. A score of 33 or higher appears reasonable to propose possible PTSD. Diagnostic criteria can also be evaluated by assessing responses to individual questions.
Depressive symptoms (adults) | 8 weeks
  Hopkins Symptoms Checklist - 25. Evaluates depressive and anxiety related symptoms in adults. Responses: ("Not at all," "A little," "Quite a bit," "Extremely," rated 1 to 4, respectively. Anxiety score is the average of the first ten questions; depressive score is the average of the last 15 questions. For either measure, scores greater than 1.75 are said to be symptomatic. Highest score = 4; lowest score = 0.
Depressive Symptoms (Children) | 8 weeks
  Mood and Feelings Questionnaire (long form). 33 questions to assess depressive symptoms, ranked from 0 to 2. Highest score = 66 and lowest = 0; score of 27 or higher is said to be indicative of possible depression. 0 = not true, 1 = sometimes true, and 2 = true.
Anxiety Symptoms (Children) | 8 weeks
  Screen for Child Anxiety Related Emotional Disorders. 41 item questionnaire. 'Not True or Hardly Ever True' (Score 0), 'Somewhat True or Sometimes True' (Score 1), or 'Very True or Often True' (Score 2). Maximum score = 82; minimum score = 0. Scores are summed.
Somatic Symptoms (adults and children) | 8 weeks
  Somatic symptoms scale, 8 items. Ranks somatic symptoms on a scale from 0 to 4, with the following possible scoring results: no to minimal (0-3 points), low (4-7 points), medium (8-11 points), high (12-15 points), and very high (16-32 points) somatic symptom burden
Inflammatory State | 8 weeks
  measure via saliva or blood
Cortisol | 8 weeks
  measure via hair

CONTACTS AND LOCATIONS:
Overall Officials: Arash Javanbakht, MD, Principal Investigator — Department of Psychiatry and Behavioral Neuroscience, Wayne State University
Locations (1):
- Wayne State U Department of Psychiatry, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grasser LR, Al-Saghir H, Wanna C, Spinei J, Javanbakht A. Moving Through the Trauma: Dance/Movement Therapy as a Somatic-Based Intervention for Addressing Trauma and Stress Among Syrian Refugee Children. J Am Acad Child Adolesc Psychiatry. 2019 Nov;58(11):1124-1126. doi: 10.1016/j.jaac.2019.07.007. Epub 2019 Jul 23. PMID 31348987